CLINICAL TRIAL: NCT01490229
Title: Randomized Trial of Ezetimibe Versus nutraCeuticals in Statin-intoLerant patIents Treated With PercutaneouS Coronary Intervention
Brief Title: Ezetimibe Versus Nutraceuticals in Statin-intolerant Patients
Acronym: ECLIPSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 651/2011/D
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: nutraceuticals; statin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ezetimibe; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Active Comparator): Patients assigned to ezetimibe will receive for 1 year ezetimibe (10 mg/day)
  Interventions: Drug: Ezetimibe
- Nutraceuticals (Active Comparator): Patients assigned to nutraceuticals will receive for 1 year 1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg
  Interventions: Drug: Nutraceuticals

INTERVENTIONS:
Drug: Ezetimibe — os, 10 mg, once daily, 1 year
  Other Names: Zetia ®, Merck, USA
  Arms: Ezetimibe
Drug: Nutraceuticals — os, 1 pill containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg, once daily, 1 year
  Other Names: Armolipid Plus, Rottapharm Madaus, Italy
  Arms: Nutraceuticals

SUMMARY:
Pharmacologic alternatives in statin-intolerant patients include ezetimibe and nutraceuticals (i.e. compounds derived from foods with cholesterol lowering actions). The investigators will compare the efficacy and tolerability of ezetimibe versus a nutraceutical-based protocol in statin-intolerant patients treated with percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background

Treatment with statins has a class I indication after percutaneous coronary intervention (PCI), but is often discontinued by patients due to side effects.

Pharmacologic alternatives shown to be useful after PCI include ezetimibe and nutraceuticals (i.e. compounds derived from foods with cholesterol lowering actions).

It remains unknown, however, which of these two therapeutic approaches is more effective after PCI.

Purpose

The primary objective of this study is to compare the efficacy and tolerability of ezetimibe versus a nutraceutical-based protocol in statin-intolerant patients treated with percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Recent (< 12 months) percutaneous coronary intervention
* Class I indication to receive statin treatment
* Previous (< 12 months) withdrawn of a statin due to side effects
* Unwilling to receive treatment with an alternative statin
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment tolerability | Up to 12 months
  Reasons for treatment discontinuation

SECONDARY OUTCOMES:
Evaluation of drug effects on lipid and metabolic features | Up to 12 months
  Effects on lipid profile (total cholesterol, LDL cholesterol, tryglicerides) and metabolic indexes (glucose levels, HOMA)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Pisana, Rome, Italy